CLINICAL TRIAL: NCT02195583
Title: The Effect of Experimental Dentifrices on Remineralization of Caries Lesions In-situ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202194; RH02437 (Other: GSK)
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-03

CONDITIONS: Oral Hygiene
MeSH Terms: interventions — Sodium Fluoride; Fluorides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sodium fluoride (1426 ppm) (Experimental): Non-zinc, 1426ppm fluoride as sodium fluoride in a silica gel base
  Interventions: Drug: Sodium fluoride (1426 ppm)
- Sodium fluoride (1150 ppm) (Experimental): Non-zinc, 1150ppm fluoride as sodium fluoride in a silica gel base
  Interventions: Drug: Sodium fluoride (1150 ppm)
- Sodium fluoride (250 ppm) (Experimental): Non-zinc, 250ppm fluoride as sodium fluoride in a silica gel base
  Interventions: Drug: Sodium fluoride (250 ppm)
- Sodium fluoride (1426 ppm) + zinc base A (Experimental): Zinc base A, 1426ppm fluoride as sodium fluoride in a silica gel base
  Interventions: Drug: Sodium fluoride (1426 ppm) + zinc base A
- Sodium fluoride (1426 ppm) + zinc base B (Experimental): Zinc base B, 1426ppm fluoride as sodium fluoride in a silica gel base
  Interventions: Drug: Sodium fluoride (1426 ppm) + zinc base B
- Fluoride (0 ppm) (Placebo Comparator): Non-zinc, 0ppm fluoride in a silica gel base
  Interventions: Drug: Fluoride (0 ppm)

INTERVENTIONS:
Drug: Sodium fluoride (1426 ppm) — Non-zinc, 1426ppm fluoride as sodium fluoride in a silica gel base
  Arms: Sodium fluoride (1426 ppm)
Drug: Sodium fluoride (1150 ppm) — Non-zinc, 1150ppm fluoride as sodium fluoride in a silica gel base
  Arms: Sodium fluoride (1150 ppm)
Drug: Sodium fluoride (250 ppm) — Non-zinc, 250ppm fluoride as sodium fluoride in a silica gel base
  Arms: Sodium fluoride (250 ppm)
Drug: Sodium fluoride (1426 ppm) + zinc base A — Zinc base A, 1426ppm fluoride as sodium fluoride in a silica gel base
  Arms: Sodium fluoride (1426 ppm) + zinc base A
Drug: Sodium fluoride (1426 ppm) + zinc base B — Zinc base B, 1426ppm fluoride as sodium fluoride in a silica gel base
  Arms: Sodium fluoride (1426 ppm) + zinc base B
Drug: Fluoride (0 ppm) — Non-zinc, 0ppm fluoride in a silica gel base
  Arms: Fluoride (0 ppm)

SUMMARY:
This study will evaluate the effect of experimental sodium fluoride-silica dentifrice formulations, with and without zinc, on remineralization of enamel in situ. Following the remineralization phase, the acid resistance of the new mineral formed will be assessed. Fluoride uptake during the remineralization phase will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Good general health with no clinically significant and relevant abnormalities of medical history or oral examination
* Participants with maxillary dental arch suitable for the retention of the palatal appliance

Exclusion Criteria:

* Participants taking fluoride supplement
* Pregnant or breast-feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one clinical study site in the USA.
Pre-assignment Details: A total of 64 participants were screened and 62 were randomized.
Groups:
- Overall Participants: Participants brushed the buccal surface of their teeth with 1.5 g (± 0.1 g) dentifrice for 25 seconds (sec) to create dentifrice slurry. Then swished the slurry around the palatal appliance for 1 minute (min) and 35 sec. Next, they expectorated the slurry, rinsed with 15 milliliter (mL) of tap water for 10 sec and expectorated. There was a 2 day washout period before each treatment period when participants used a non-fluoridated dentifrice.
  1. Sodium fluoride (1426 ppm):Non-zinc, 1426ppm fluoride as sodium fluoride in silica base
  2. Sodium fluoride (1150 ppm):Non-zinc, 1150ppm fluoride as sodium fluoride in silica base
  3. Sodium fluoride (250 ppm):Non-zinc, 250ppm fluoride as sodium fluoride in silica base
  4. Sodium fluoride (1426 ppm) + zinc base A:Zinc base A, 1426ppm fluoride as sodium fluoride in silica base
  5. Sodium fluoride (1426 ppm) + zinc base B:Zinc base B, 1426ppm fluoride as sodium fluoride in silica base
  6. Sodium fluoride (0 ppm):Non-zinc, 0ppm fluoride in silica base
Period: Overall Study
Arm/Group | Overall Participants
Started | 62
Sodium Fluoride (1150 Ppm) | 57 (Discontinuations: 1 due to other reason in Period 5)
Sodium Fluoride (0 Ppm) | 59
Sodium Fluoride (1426 Ppm) + Zinc Base A | 58 (Discontinuations: 1 withdrawal of consent in Period 3 and 1 withdrawal of consent in Period 4)
Sodium Fluoride (250 Ppm) | 55
Sodium Fluoride (1426 Ppm) | 59 (Discontinuation:1 lost to follow up, 1 withdrawal of consent in Period 2, 1 other reason in Period 5)
Sodium Fluoride (1426 Ppm) + Zinc Base B | 60 (Discontinuations: 1 withdrawal of consent in Period 2;1 adverse event each in Period 3 and Period 4)
Completed | 53
Not Completed | 9
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 2
Not completed — Other Reason | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants were evaluated for baseline characteristics
Groups:
- All Randomized Participants: All randomized participants were evaluated for baseline characteristics
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage Surface Microhardness Recovery (% SMHR)
Description: Changes in the mineral content of the four centrally-located enamel specimens were evaluated using the Surface Microhardness (SMH) Test. The SMH was measured using a Wilson 2100 Hardness Tester. The baseline SMH was determined prior to the in vitro acid challenge. SMH was determined again after the in vitro acid challenge, after the in situ remineralization test, and again after the second in vitro acid challenge. The extent of remineralization was calculated as the % recovery in SMH using the equation: % SMHR= [(D1-R)/(D1-B)]*100 Where B = indentation length (μm) of sound enamel at baseline; D1 = indentation length (μm) after first acid challenge; R = indentation length (μm) after in situ remineralization.
Time Frame: Baseline to 4 hours
Population: The primary population for the efficacy analysis was the Per Protocol (PP) population, including participants with a protocol violation affecting some (but not all) of the efficacy assessments. However, data from assessments when a violation occurred were excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of SMHR
Groups:
- Sodium Fluoride (1426 Ppm): Non-zinc, 1426ppm fluoride as sodium fluoride in a silica base. Participants brushed the buccal surface of their teeth with 1.5 g (± 0.1 g) dentifrice for 25 sec to create dentifrice slurry. Next, they swished the dentifrice slurry around the palatal appliance for 1 min and 35 sec. After that, participants expectorated the slurry, gently but thoroughly rinsed with 15 mL of tap water for 10 sec and expectorated again. There was a 2 day wash-out period before each treatment period when participants used a non-fluoridated dentifrice.
- Sodium Fluoride (1150 Ppm): Non-zinc, 1150ppm fluoride as sodium fluoride in a silica base. Participants brushed the buccal surface of their teeth with 1.5 g (± 0.1 g) dentifrice for 25 sec to create dentifrice slurry. Next, they swished the dentifrice slurry around the palatal appliance for 1 min and 35 sec. After that, participants expectorated the slurry, gently but thoroughly rinsed with 15 mL of tap water for 10 sec and expectorated again. There was a 2 day wash-out period before each treatment period when participants used a non-fluoridated dentifrice.
- Sodium Fluoride (250 Ppm): Non-zinc, 250ppm fluoride as sodium fluoride in a silica base. Participants brushed the buccal surface of their teeth with 1.5 g (± 0.1 g) dentifrice for 25 sec to create dentifrice slurry. Next, they swished the dentifrice slurry around the palatal appliance for 1 min and 35 sec. After that, participants expectorated the slurry, gently but thoroughly rinsed with 15 mL of tap water for 10 sec and expectorated again. There was a 2 day wash-out period before each treatment period when participants used a non-fluoridated dentifrice.
- Sodium Fluoride (1426 Ppm) + Zinc Base A: Zinc base A, 1426ppm fluoride as sodium fluoride in a silica base. Participants brushed the buccal surface of their teeth with 1.5 g (± 0.1 g) dentifrice for 25 sec to create dentifrice slurry. Next, they swished the dentifrice slurry around the palatal appliance for 1 min and 35 sec. After that, participants expectorated the slurry, gently but thoroughly rinsed with 15 mL of tap water for 10 sec and expectorated again. There was a 2 day wash-out period before each treatment period when participants used a non-fluoridated dentifrice.
- Sodium Fluoride (1426 Ppm) + Zinc Base B: Zinc base B, 1426ppm fluoride as sodium fluoride in a silica base. Participants brushed the buccal surface of their teeth with 1.5 g (± 0.1 g) dentifrice for 25 sec to create dentifrice slurry. Next, they swished the dentifrice slurry around the palatal appliance for 1 min and 35 sec. After that, participants expectorated the slurry, gently but thoroughly rinsed with 15 mL of tap water for 10 sec and expectorated again. There was a 2 day wash-out period before each treatment period when participants used a non-fluoridated dentifrice.
- Sodium Fluoride (0 Ppm): Non-zinc, 0ppm fluoride in a silica base. Participants brushed the buccal surface of their teeth with 1.5 g (± 0.1 g) dentifrice for 25 sec to create dentifrice slurry. Next, they swished the dentifrice slurry around the palatal appliance for 1 min and 35 sec. After that, participants expectorated the slurry, gently but thoroughly rinsed with 15 mL of tap water for 10 sec and expectorated again. There was a 2 day wash-out period before each treatment period when participants used a non-fluoridated dentifrice.
Arm/Group | Sodium Fluoride (1426 Ppm) | Sodium Fluoride (1150 Ppm) | Sodium Fluoride (250 Ppm) | Sodium Fluoride (1426 Ppm) + Zinc Base A | Sodium Fluoride (1426 Ppm) + Zinc Base B | Sodium Fluoride (0 Ppm)
Number analyzed (Participants) | 59 | 57 | 55 | 58 | 60 | 59
Percentage of SMHR | 32.49 (1.167) | 31.81 (1.182) | 27.56 (1.199) | 22.62 (1.175) | 23.22 (1.159) | 24.78 (1.167)
Statistical Analysis 1: Comparison: Sodium Fluoride (1426 Ppm) vs Sodium Fluoride (1150 Ppm) vs Sodium Fluoride (250 Ppm); Linear contrasts were fitted in order to establish whether there was a dose-response relationship. Linear contrasts were for experimental dentifrice: non-zinc treatments; Test type: Superiority or Other; p < 0.0001, ANOVA; Calculated from Analysis of Variance (ANOVA) model using treatment and study period as fixed factors and participant as random effect
Statistical Analysis 2: Comparison: Sodium Fluoride (1426 Ppm) vs Sodium Fluoride (1150 Ppm) vs Sodium Fluoride (250 Ppm); Quadratic contrasts were fitted in order to establish whether there was a dose-response relationship. Quadratic contrasts are for experimental dentifrice: non-zinc treatments; Test type: Superiority or Other; p = 0.2274, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect
Statistical Analysis 3: Comparison: Sodium Fluoride (1426 Ppm) vs Sodium Fluoride (1150 Ppm); Test type: Superiority or Other; p = 0.5950, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect; Mean Difference (Net) = 0.68, 95% CI 2-sided [-1.84 to 3.20] — Difference was calculated as Sodium fluoride (1426 ppm) minus Sodium fluoride (1150 ppm) such that a positive difference favors Sodium fluoride (1426 ppm)
Statistical Analysis 4: Comparison: Sodium Fluoride (1426 Ppm) vs Sodium Fluoride (250 Ppm); Test type: Superiority or Other; p = 0.0002, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect; Mean Difference (Net) = 4.93, 95% CI 2-sided [2.38 to 7.48] — Difference was calculated as Sodium fluoride (1426 ppm) minus Sodium fluoride (250 ppm) such that a positive difference favors Sodium fluoride (1426 ppm)
Statistical Analysis 5: Comparison: Sodium Fluoride (1150 Ppm) vs Sodium Fluoride (250 Ppm); Test type: Superiority or Other; p = 0.0013, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect; Mean Difference (Net) = 4.25, 95% CI 2-sided [1.68 to 6.82] — Difference was calculated as Sodium fluoride (1150 ppm) minus Sodium fluoride (250 ppm) such that a positive difference favors Sodium fluoride (1150 ppm)
Statistical Analysis 6: Comparison: Sodium Fluoride (1426 Ppm) vs Sodium Fluoride (0 Ppm); Test type: Superiority or Other; p < 0.0001, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect; Mean Difference (Net) = 7.71, 95% CI 2-sided [5.20 to 10.21] — Difference was calculated as Sodium fluoride (1426 ppm) minus Sodium fluoride (0 ppm) such that a positive difference favors Sodium fluoride (1426 ppm)
Statistical Analysis 7: Comparison: Sodium Fluoride (1150 Ppm) vs Sodium Fluoride (0 Ppm); Test type: Superiority or Other; p < 0.0001, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect; Mean Difference (Net) = 7.03, 95% CI 2-sided [4.51 to 9.55] — Difference was calculated as Sodium fluoride (1150 ppm) minus Sodium fluoride (0 ppm) such that a positive difference favors Sodium fluoride (1150 ppm)
Statistical Analysis 8: Comparison: Sodium Fluoride (250 Ppm) vs Sodium Fluoride (0 Ppm); Test type: Superiority or Other; p = 0.0325, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect; Mean Difference (Net) = 2.78, 95% CI 2-sided [0.23 to 5.32] — Difference was calculated as Sodium fluoride (250 ppm) minus Sodium fluoride (0 ppm) such that a positive difference favors Sodium fluoride (250 ppm)
Statistical Analysis 9: Comparison: Sodium Fluoride (1426 Ppm) + Zinc Base A vs Sodium Fluoride (0 Ppm); Test type: Superiority or Other; p = 0.0920, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect; Mean Difference (Net) = -2.16, 95% CI 2-sided [-4.67 to 0.35] — Difference was calculated as 'Sodium fluoride (1426 ppm) + zinc base A' minus Sodium fluoride (0 ppm) such that a positive difference favors 'Sodium fluoride (1426 ppm) + zinc base A'
Statistical Analysis 10: Comparison: Sodium Fluoride (1426 Ppm) + Zinc Base B vs Sodium Fluoride (0 Ppm); Test type: Superiority or Other; p = 0.2185, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect; Mean Difference (Net) = -1.56, 95% CI 2-sided [-4.04 to 0.93] — Difference was calculated as 'Sodium fluoride (1426 ppm) + zinc base B' minus Sodium fluoride (0 ppm) such that a positive difference favors 'Sodium fluoride (1426 ppm) + zinc base B'
Statistical Analysis 11: Comparison: Sodium Fluoride (1426 Ppm) vs Sodium Fluoride (1426 Ppm) + Zinc Base A; Test type: Superiority or Other; p < 0.0001, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect; Mean Difference (Net) = 9.87, 95% CI 2-sided [7.36 to 12.37] — Difference was calculated as Sodium fluoride (1426 ppm) minus 'Sodium fluoride (1426 ppm) + zinc base A' such that a positive difference favors Sodium fluoride (1426 ppm)
Statistical Analysis 12: Comparison: Sodium Fluoride (1426 Ppm) vs Sodium Fluoride (1426 Ppm) + Zinc Base B; Test type: Superiority or Other; p < 0.0001, ANOVA; Calculated from ANOVA model using treatment and study period as fixed factors and participant as random effect; Mean Difference (Net) = 9.26, 95% CI 2-sided [6.77 to 11.75] — Difference was calculated as Sodium fluoride (1426 ppm) minus 'Sodium fluoride (1426ppm) + zinc base B' such that a positive difference favors Sodium fluoride (1426 ppm)

2. Secondary Outcome: Enamel Fluoride Uptake
Description: The microdrill enamel biopsy technique was used to analyze the fluoride uptake by enamel. Each enamel specimen was mounted on the long axis of a drill attached to a microdrill and drilled to a depth of approximately 100 micrometer (μm) through the entire lesion (four cores per specimen). The enamel powder pooled from four drilling sample was then immediately analyzed for fluoride content using fluoride specific electrode and pH/ion meter. The amount of fluoride-uptake by enamel was calculated based on the amount of fluoride divided by the area of the enamel cores and expressed as microgram per square centimeter (μg/cm^2).
Time Frame: Baseline to 4 hours
Population: The main population for the secondary efficacy analysis was the PP population, including participants with a protocol violation affecting some (but not all) of the efficacy assessments. However, data from assessments when a violation occurred were excluded.
Measure: Least Squares Mean (Standard Error); unit: microgram per square centimeter(μg/cm^2)
Arm/Group | Sodium Fluoride (1426 Ppm) | Sodium Fluoride (1150 Ppm) | Sodium Fluoride (250 Ppm) | Sodium Fluoride (1426 Ppm) + Zinc Base A | Sodium Fluoride (1426 Ppm) + Zinc Base B | Sodium Fluoride (0 Ppm)
Number analyzed (Participants) | 59 | 57 | 55 | 58 | 60 | 59
microgram per square centimeter(μg/cm^2) | 2.94 (0.083) | 2.70 (0.084) | 1.85 (0.085) | 2.62 (0.083) | 2.37 (0.082) | 0.98 (0.083)

3. Secondary Outcome: Percentage Net Acid Resistance (% NAR)
Description: Changes in the mineral content of the four centrally-located enamel specimens were evaluated using the SMH Test. The SMH was measured using a Wilson 2100 Hardness Tester. The baseline SMH was measured prior to the in vitro acid challenge. SMH was measured again after the in vitro acid challenge, after the in situ remineralization test, and again after the second in vitro acid challenge. The % NAR was calculated using the equation: % NAR= [(D1-D2)/(D1-B)]*100 where B= Indentation length (μm) of sound enamel at baseline; D1= Indentation length (μm) after first acid challenge and D2= Indentation length (μm) after second acid challenge.
Time Frame: Baseline to 4 hours
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of NAR
Arm/Group | Sodium Fluoride (1426 Ppm) | Sodium Fluoride (1150 Ppm) | Sodium Fluoride (250 Ppm) | Sodium Fluoride (1426 Ppm) + Zinc Base A | Sodium Fluoride (1426 Ppm) + Zinc Base B | Sodium Fluoride (0 Ppm)
Number analyzed (Participants) | 59 | 57 | 55 | 58 | 60 | 59
Percentage of NAR | -12.54 (1.224) | -13.45 (1.244) | -17.81 (1.266) | -17.60 (1.234) | -18.98 (1.214) | -50.60 (1.224)

4. Secondary Outcome: Percentage Comparative Acid Resistance (% CAR)
Description: Changes in the mineral content of the four centrally-located enamel specimens were evaluated using the SMH Test. The SMH was measured using a Wilson 2100 Hardness Tester. The baseline SMH was measured prior to the in vitro acid challenge. SMH was measured again after the in vitro acid challenge, after the in situ remineralization test, and again after the second in vitro acid challenge. The % CAR was calculated using the equation: % CAR= [(D2-R)/(D1-B)]*100 where B= Indentation length (μm) of sound enamel at baseline; R= Indentation length (μm) of enamel after in situ remineralization; D1= Indentation length (μm) after first acid challenge; D2= Indentation length (μm) after second acid challenge.
Time Frame: Baseline to 4 hours
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of CAR
Groups:
- Sodium Fluoride (0 Ppm): Sodium fluoride (0 ppm) Non-zinc, 0ppm fluoride in a silica base. Participants brushed the buccal surface of their teeth with 1.5 g (± 0.1 g) dentifrice for 25 sec to create dentifrice slurry. Next, they swished the dentifrice slurry around the palatal appliance for 1 min and 35 sec. After that, participants expectorated the slurry, gently but thoroughly rinsed with 15 mL of tap water for 10 sec and expectorated again. There was a 2 day wash-out period before each treatment period when participants used a non-fluoridated dentifrice.
Arm/Group | Sodium Fluoride (1426 Ppm) | Sodium Fluoride (1150 Ppm) | Sodium Fluoride (250 Ppm) | Sodium Fluoride (1426 Ppm) + Zinc Base A | Sodium Fluoride (1426 Ppm) + Zinc Base B | Sodium Fluoride (0 Ppm)
Number analyzed (Participants) | 59 | 57 | 55 | 58 | 60 | 59
Percentage of CAR | 45.00 (1.274) | 45.23 (1.295) | 45.44 (1.319) | 40.29 (1.285) | 42.21 (1.264) | 75.41 (1.274)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the start of the investigational product (or washout product) and until five days following last administration of the investigational product.Serious adverse events (SAEs) were collected over the same time period.
Arm/Group | Sodium Fluoride (1426 Ppm) | Sodium Fluoride (1150 Ppm) | Sodium Fluoride (250 Ppm) | Sodium Fluoride (1426 Ppm) + Zinc Base A | Sodium Fluoride (1426 Ppm) + Zinc Base B | Sodium Fluoride (0 Ppm)
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/57 | 0/55 | 0/58 | 1/60 | 0/59
Other Adverse Events (participants affected / at risk) | 3/59 | 1/57 | 5/55 | 1/58 | 4/60 | 5/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Fluoride (1426 Ppm) (N=59) | Sodium Fluoride (1150 Ppm) (N=57) | Sodium Fluoride (250 Ppm) (N=55) | Sodium Fluoride (1426 Ppm) + Zinc Base A (N=58) | Sodium Fluoride (1426 Ppm) + Zinc Base B (N=60) | Sodium Fluoride (0 Ppm) (N=59)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Fluoride (1426 Ppm) (N=59) | Sodium Fluoride (1150 Ppm) (N=57) | Sodium Fluoride (250 Ppm) (N=55) | Sodium Fluoride (1426 Ppm) + Zinc Base A (N=58) | Sodium Fluoride (1426 Ppm) + Zinc Base B (N=60) | Sodium Fluoride (0 Ppm) (N=59)
Oral Mucosal Erythema (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Parotid Gland Enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1
Lymph gland infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.